CLINICAL TRIAL: NCT00398216
Title: A Phase IIb, Randomized, Parallel Group, Double-Blind, Double-Dummy, Multi-Center, Multi-National, Multi-Dose, Study of DU-176b Compared to Dalteparin in Patients Undergoing Elective Unilateral Total Hip Replacement
Brief Title: A Study of DU-176b in Preventing Blood Clots After Hip Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Anne MacDonald, Daiichi Sankyo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DU176b-PRT011; 2006-000758-29 (EudraCT Number)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2015-02-25 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2015-02

CONDITIONS: Thrombosis; Hip Replacement
Keywords: Anti-coagulant; hip replacement; hip replacement surgery; unilateral hip replacement surgery; DeepVein Thrombosis; Venous Thromboembolism; pulmonary embolism; Prevention of Blood Clots
MeSH Terms: conditions — Thrombosis; Venous Thromboembolism; Pulmonary Embolism

INTERVENTIONS:
Drug: DU176b - action is the prevention of venous thromboembolism by the use of a Factor Xa inhibitor

SUMMARY:
This study is to assess if DU176b is effective in prevention of blood clots following hip replacement surgery. The duration is 7-10 days of treatment and 30 and 60 day follow-up visits.

ELIGIBILITY:
1. 18 years of age or older; male or female.
2. Able to provide written informed consent.
3. Must be scheduled for elective unilateral total hip replacement surgery. Only primary surgeries accepted.
4. If female, must be either one year post-menopausal, surgically sterile, or using medically accepted contraceptive measures as judged by the Investigator and in accordance with local regulatory requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (3):
  - Hartford, Connecticut
  - Sarasota, Florida
  - Austin, Texas
- Canada (5):
  - Ajax, Ontario
  - Cambridge, Ontario
  - Guelph, Ontario
  - Kitchner, Ontario
  - Toronto, Ontario
- Denmark (3):
  - Hellerup
  - Herlev
  - Hørsholm
- Hungary (3):
  - Gyula
  - Kecskemét
  - Szeged
- Riga, Latvia
- Russia (6):
  - Krasnoyarsk
  - Moscow
  - Saint Petersburg
  - Saratov
  - Veliky Novgorod
  - Volgograd
- Ukraine (8):
  - Chernivtsy
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kiev
  - Lutsk
  - Lviv
  - Odesa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Groups:
- Edoxaban 15mg QD: edoxaban 15mg QD (once daily) orally (PO)
- Edoxaban 30mg QD: edoxaban 30mg QD PO
- Edoxaban 60mg QD: edoxaban 60mg QD PO
- Edoxaban 90mg QD: edoxaban 90mg QD PO
- Dalteparin: dalteparin 2500 IU/mL initial dose followed by 5000 IU once daily subcutaneously
Period: Overall Study
Arm/Group | Edoxaban 15mg QD | Edoxaban 30mg QD | Edoxaban 60mg QD | Edoxaban 90mg QD | Dalteparin
Started | 192 | 170 | 185 | 177 | 172
Completed | 181 | 151 | 164 | 155 | 157
Not Completed | 11 | 19 | 21 | 22 | 15
Not completed — Adverse Event | 4 | 2 | 5 | 7 | 2
Not completed — Protocol Violation | 2 | 4 | 5 | 7 | 5
Not completed — Lost to Follow-up | 1 | 6 | 4 | 4 | 1
Not completed — Death | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 1 | 2
Not completed — administrative reasons | 3 | 4 | 4 | 3 | 3
Not completed — entrance criteria | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban 15mg QD | Edoxaban 30mg QD | Edoxaban 60mg QD | Edoxaban 90mg QD | Dalteparin | Total
Number analyzed (Participants) | 192 | 170 | 185 | 177 | 172 | 896
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 126 | 111 | 126 | 114 | 110 | 587
  >=65 years | 66 | 59 | 59 | 63 | 62 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.49) | 57.2 (12.28) | 58.3 (11.52) | 58.5 (12.27) | 57.5 (12.43) | 57.8 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 111 | 118 | 93 | 105 | 540
  Male | 79 | 59 | 67 | 84 | 67 | 356
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 1 | 4 | 10
  White | 188 | 167 | 178 | 176 | 165 | 874
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3 | 0 | 3 | 9
Region of Enrollment [Number; unit: participants]
  North America | 33 | 20 | 33 | 33 | 29 | 148
  Europe | 159 | 150 | 152 | 144 | 143 | 748

OUTCOME MEASURES:

1. Primary Outcome: Adjudicated Incidence of VTE
Description: Assess the efficacy of DU-176b in the prevention of venous thromboembolism (VTE) from 6 to 8 hours after hip replacement surgery to 7 to 10 days after the surgery.
  A subject was judged to have a VTE if one or more of the following criteria were met:
  * Observed lower extremity deep vein thrombosis (DVT) (either proximal, distal, or both ) as assessed by bilateral or unilateral ascending contrast venography prior to or at the end-of-treatment (EOT) visit
  * Symptomatic and objectively proven pulmonary embolism prior to or at the EOT visit
  * Symptomatic and objectively proven DVT prior to or at EOT visit end of treatment defined as 6 to 8 hours after after hip replacement surgery to 7 to 10 days after the surgery.
Time Frame: end of treatment
Population: per protocol analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants with VTE
Arm/Group | Edoxaban 15mg QD | Edoxaban 30mg QD | Edoxaban 60mg QD | Edoxaban 90mg QD | Dalteparin
Number analyzed (Participants) | 162 | 143 | 153 | 139 | 137
percentage of participants with VTE | 29.0 [22.2 to 36.7] | 20.3 [14.0 to 27.8] | 15.7 [10.3 to 22.4] | 11.5 [6.7 to 18.0] | 46.0 [37.4 to 54.7]
Statistical Analysis 1: Comparison: Edoxaban 15mg QD vs Dalteparin; Test type: Superiority or Other; p = 0.003, Fisher Exact
Statistical Analysis 2: Comparison: Edoxaban 30mg QD vs Dalteparin; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Edoxaban 60mg QD vs Dalteparin; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Edoxaban 90mg QD vs Dalteparin; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Change in Prothrombin Time (PT) From Baseline
Description: change in prothrombin time (PT) from baseline to end of treatment end of treatment defined as 6-8 hours after hip replacement surgery to 7 to 10 days after the surgery
Time Frame: end of treatment
Population: perp protocol analysis set
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Edoxaban 15mg QD | Edoxaban 30mg QD | Edoxaban 60mg QD | Edoxaban 90mg QD | Dalteparin
Number analyzed (Participants) | 153 | 137 | 146 | 134 | 132
seconds | .90 (3.205) | 1.07 (1.875) | 2.87 (6.279) | 2.74 (5.821) | .67 (1.88)

3. Secondary Outcome: Change in Activated Partial Thromboplastin Time (aPTT) From Baseline
Description: change in Activated Partial Thromboplastin Time (aPTT) from baseline to end of treatment end of treatment defined as 6-8 hours after hip replacement surgery to 7 to 10 days after the surgery
Time Frame: end of treatment
Population: perp protocol analysis set
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Edoxaban 15mg QD | Edoxaban 30mg QD | Edoxaban 60mg QD | Edoxaban 90mg QD | Dalteparin
Number analyzed (Participants) | 149 | 137 | 145 | 134 | 131
seconds | -0.33 (6.562) | 1.67 (13.092) | 4.39 (16.930) | 3.26 (13.169) | 2.34 (12.396)

4. Secondary Outcome: Adjudicated Incidence of Major or Clinically Relevant Non-major Bleeding Events
Description: adjudicated incidence of major or clinically relevant non-major bleeding events through 10 days after first dose
Time Frame: 10 days after first dose
Population: safety analysis dataset
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleed events
Arm/Group | Edoxaban 15mg QD | Edoxaban 30mg QD | Edoxaban 60mg QD | Edoxaban 90mg QD | Dalteparin
Number analyzed (Participants) | 192 | 170 | 185 | 177 | 172
percentage of subjects with bleed events | 1.6 [0.3 to 4.5] | 1.8 [0.4 to 5.1] | 2.2 [0.6 to 5.4] | 2.3 [0.6 to 5.7] | 0 [0.0 to 2.1]
Statistical Analysis 1: Comparison: Edoxaban 15mg QD vs Dalteparin; Test type: Superiority or Other; p = .250, Fisher Exact
Statistical Analysis 2: Comparison: Edoxaban 30mg QD vs Dalteparin; Test type: Superiority or Other; p = .122, Fisher Exact
Statistical Analysis 3: Comparison: Edoxaban 60mg QD vs Dalteparin; Test type: Superiority or Other; p = .124, Fisher Exact
Statistical Analysis 4: Comparison: Edoxaban 90mg QD vs Dalteparin; Test type: Superiority or Other; p = .123, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Edoxaban 15mg QD | Edoxaban 30mg QD | Edoxaban 60mg QD | Edoxaban 90mg QD | Dalteparin
Serious Adverse Events (participants affected / at risk) | 8/192 | 6/170 | 8/185 | 10/177 | 3/172
Other Adverse Events (participants affected / at risk) | 30/192 | 16/170 | 22/185 | 25/177 | 22/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edoxaban 15mg QD (N=192) | Edoxaban 30mg QD (N=170) | Edoxaban 60mg QD (N=185) | Edoxaban 90mg QD (N=177) | Dalteparin (N=172)
acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
secretion of discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
fat embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
incision site hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
post-procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
cardiovascular insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
hematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
wound hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban 15mg QD (N=192) | Edoxaban 30mg QD (N=170) | Edoxaban 60mg QD (N=185) | Edoxaban 90mg QD (N=177) | Dalteparin (N=172)
constipation (Gastrointestinal disorders) | 5 | 3 | 8 | 14 | 6
nausea (Gastrointestinal disorders) | 13 | 4 | 8 | 8 | 6
edema peripheral (General disorders) | 11 | 5 | 7 | 6 | 8
pyrexia (General disorders) | 15 | 3 | 8 | 6 | 6
procedural pain (Injury, poisoning and procedural complications) | 10 | 5 | 8 | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A study site may not publish results of a study until after a coordinated multicenter publication has been submitted for publication or until one year after the study has ended, whichever occurs first. The study site will have the opportunity to publish results of the study, provided Daiichi Sankyo has had the opportunity to review and comment on the study site's proposed publication prior to being submitted for publication with the advice of patent council and need for subject protection.